CLINICAL TRIAL: NCT05404828
Title: TUCSON Study: Tackling Underlying Causes of Sleep Related Nocturia
Brief Title: TUCSON Study: Tackling Underlying Causes of Sleep Related Nocturia Nocturia
Acronym: TUCSON
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10535
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nocturia; Insomnia; OSA
Keywords: Nocturia; Insomnia; Sleep Apnea, Obstructive; Polysomnography
MeSH Terms: conditions — Nocturia; Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- OSAS: All adult patients consulting the pneumology department for possible OSAS with >1x/night nocturia
  Interventions: Other: Polysomnography; Other: Questionnaires; Other: Blood and urine sample
- Insomnia: All adult patients consulting the center for integrative medicine for insomnia with >1x/night nocturia
  Interventions: Other: Polysomnography; Other: Questionnaires; Other: Blood and urine sample
- Urological: All adult patients consulting the urology department with >1x/night nocturia
  Interventions: Other: Polysomnography; Other: Questionnaires; Other: Blood and urine sample

INTERVENTIONS:
Other: Polysomnography — Polysomnography: WASO, FUSP, TST, TIB, SEF, Global Wake Index, Sleep Latency, AHI
Other: Questionnaires — STOP-BANG, ISI, ESS, PSQI, MTCQ, ICIQ-F/MLUTS, IRLS, TANGO, SF36
Other: Blood and urine sample — Na, K, Creat, Osm, Urea

SUMMARY:
The TUCSON study is a cross-sectional observational monocentric study. In order to provide a clinical helpful assessment for urologists for possible missed causes of nocturia, the aim is to investigate the voiding and sleep pattern through questionnaires and sleep and voiding diaries of patients consulting the urology department, sleep clinic and pneumology department. An assessment of the prevalence of missed underlying causes will be made and a subset of patients will be asked to deliver urine samples from every night time and first morning void to further investigate possible differences in urine content between the groups. First of all, with this research the aim to offer an idea about the order of magnitude for missed underlying causes of nocturia. Secondly, to discover a specific sleep and voiding pattern for the different entities of nocturia and thirdly, to offer a useful screening tool for underlying pathology in clinical practice.

DETAILED DESCRIPTION:
Study rationale and unmet medical need:

In current urological practice, patients complaining from nocturia are not systematically screened for underlying pathology that could cause their nocturnal voiding complaints. Even though guidelines recommend screening for other factors besides the urological ones, it remains difficult to implement these strategies in daily practice during consultation. Clear cut questionnaires to screen for OSAS or underlying sleep disorders remain cumbersome and it is yet to be investigated if there is a difference in voiding and sleep pattern between the different causal entities of nocturia.

In order to provide a clinical helpful assessment for urologists for possible missed causes of nocturia, we aim to investigate the voiding and sleep pattern through questionnaires and sleep and voiding diaries in patients consulting the urology department, sleep clinic and pneumology department. An assessment of the prevalence of missed underlying causes will be made and a subset of patients will be asked to deliver urine samples from every night time and first morning void to further investigate possible differences in urine content between the groups.

First of all, with this research the aim is to offer an idea about the order of magnitude for missed underlying causes of nocturia. Secondly, to offer a useful screening tool for underlying pathology in clinical practice and thirdly, to discover a specific sleep and voiding pattern for the different entities of nocturia.

Study objectives:

* To gather cross-sectional information about the underlying cause of nocturia in patients consulting a urologist, sleep specialist or pneumologist.
* The collected data will be saved in a protected and pseudonymised database.
* Sleep, urinary symptoms, sleep apnea and quality of life will be assessed through appropriate questionnaires that patients will need to fill in before treatment.
* The tango questionnaire will be compared to the results from the above mentioned questionnaires in order to assess the value of the Tango questionnaire as a complete screening tool for underlying causes of nocturia, even in first line practice.
* A subset of patients will be asked to take urine samples from every night time and first void in the morning during one night, with a fasting blood collection the following morning. For patients undergoing a PSG, the urine collection and blood draw will be collected during that night.
* Patients will be asked to keep a 7 day nighttime only voiding diary, a 7 day sleep diary and a 3 day FVC. Patients undergoing a PSG will be asked to fill in the last day of their sleep and voiding diary during that night.
* Validation of the FUSP (First Uninterrupted Sleep Period) concept, by comparing data from the PSG to the sleep and voiding diaries.
* Information on comorbidities, medical history and medication use will be derived from the electronic patient files.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 years
* Nocturia 2x/night or more

Exclusion Criteria:

* current UTI
* SNM during the last year
* Botox during the last year
* working night shifts during the past 2 weeks
* Pregnant or breastfeeding women
* PTNS/SANS during the past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included by their treating physician from either the urology department for complaints of nocturia, the pneumology department for OSAS or the center for integrative medicine for insomnia complaints.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Voiding pattern | 1 week
  Differences in voiding frequency volume charts

SECONDARY OUTCOMES:
Sleep pattern | 1 week
  Differences in sleeping parameters derived from PSG and sleep diaries. The combined measurements will provide information on sleep quality, total sleep time, the number of awakenings etc
Solute excretion | 1 night
  Differences in urinary composition: Na, Urea, Osm, Creat

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Fanders, Belgium

IPD SHARING:
Plan to Share IPD: No